CLINICAL TRIAL: NCT04327414
Title: The Effect of Standing Desks in Secondary Schools on Sedentary Behavior and Cognitive Performance in Flemish Adolescents
Brief Title: The Effect of Standing Desks on Cognitive Performance in Adolescents
Acronym: UP4BRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UP4BRAINS
Record Dates: First submitted 2020-03-11; First posted 2020-03-31 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-03

CONDITIONS: Sedentary Behavior
Keywords: Adolescent; Classroom; Standing desk; Sitting; Standing; Cognition; Cognitive function; Cognitive performance; Sleep; Sleep quality; Sleep duration
MeSH Terms: conditions — Sedentary Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Controlled trial:
  December-January 2020: Recruitment of six secondary schools with immediate allocation to the intervention or control condition and collecting informed consents.
  February 2020: Pre-test data collection, installing standing desks in intervention schools.
  March 2020: Interruption of the study due to COVID-19 pandemic. September-October 2020: Recruitment of six new classes and collecting informed consents, pre-test data collection.
  November-December 2020: Post-test data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implementation of standing desks in classroom. To ensure that adolescents will spend sufficient time at the standing desks, 1/3 to half of the classroom will be provided with standing desks. The school will be asked to actually replace some traditional desks with these standing desks, instead of just adding standing desks to the classroom set-up to ensure as much as possible that the desks are being continuously used throughout the intervention period.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): No implementation of standing desks in classroom.

INTERVENTIONS:
Behavioral: Intervention group — Standing desks
  Arms: Intervention group

SUMMARY:
Sitting or sedentary behavior is associated with several adverse health outcomes such as overweight and obesity, diabetes type 2,... independent of physical activity levels. This evidence is clear in adults, however also in adolescents the health effects can become apparent (e.g. development of overweight, reduced fitness,...). Therefore it is important to develop interventions aiming to reduce sedentary behavior in adolescents. Adolescents are sedentary for more than 60% of the day, of wich a large part is spent at school as during school hours pupils usually have to sit at their desk. Therefore secondary schools serve as an ideal setting to target sitting behavior. Structural environmental changes (in the classroom), e.g. introducing standing desks, can be used as a possible strategy.

It is important to objectively evaluate the effect of the intervention on sedentary behavior. Next to evaluating the effect on behavior, studies also recommend to evaluate the effect on cognitive performance, as this is the particular interest of schools and their staff.

The primary aim of this project is therefore to investigate the effect of implementing standing desks on adolescents' cognitive function, more specifically on memory, reasoning, verbal ability and concentration. In addition, the investigators will evaluate the effect of implementing standing desks on adolescents' sitting and standing time, measured by Axivity accelerometers in the entire sample. Finally, the investigators will also collect information about sleeping behavior to investigate the association with cognitive performance. This will be tested via a controlled trial with a pre- and post-test design including an intervention and control group. Based on previous research studies, the hypothesis is that adolescents from the intervention group will improve their cognitive function and standing time and reduce their sitting time, whereas no changes are expected to be found for adolescents from the control group. Finally, it is expected that a more healthy sleeping behavior is associated with better cognitive performance.

DETAILED DESCRIPTION:
Introduction:

Sedentary behavior is defined as "any waking behavior characterized by an energy expenditure ≤1.5 metabolic equivalents (METs), while in a sitting, reclining or lying posture". Among adults, evidence suggests that prolonged time spent in sedentary behavior is positively associated with type 2 diabetes, cardiovascular diseases, metabolic syndrome and all-cause mortality. Although this association is less consistent among children and adolescents, several studies and reviews have found adverse associations between sedentary time and health outcomes in children and adolescents too. Additionally, a review of reviews has found evidence for an association between screen-time behaviors (i.e. specific sedentary behaviors) and obesity and moderate evidence for an association between screen-time behaviors and blood pressure, total cholesterol, self-esteem, social behavior problems, physical fitness and academic achievement, and these associations are largely independent from moderate- to vigorous physical activity. Moreover, since sedentary time in early life tracks into adulthood where it can have potential health implications, strategies are needed to reduce sedentary time in children and adolescents. Children and adolescents spend more than 60% of the day (waking hours) sedentary. In addition, more than 65% of the time at school is spent in sedentary activities. Therefore, the classroom can be considered an important setting for implementing specific strategies to reduce sedentary time in this target group.

A potential environmental strategy to reduce sedentary time during school hours is replacing traditional desks and chairs with standing desks. Although there is currently no general consensus on the health benefits of implementing standing desks into the classroom, this strategy might have a beneficial impact on children's energy expenditure. For sedentary time, standing time and step counts, results are currently mixed. More research is needed to make strong conclusions, as previous studies often had a low quality design. Furthermore, it is also advocated to focus on secondary schoolchildren, as the majority of studies have been conducted in primary schools and the level of sedentary behavior is high in secondary schools.

However, qualitative data from teachers in secondary schools from a study conducted previously by our research group (see references) indicated that not all teachers are convinced of the added value of implementing standing desks in secondary schools. The major worry is that standing up during lessons might impact pupils' academic performance. As this is a genuine concern, robust evidence that standing desks have positive effects on pupils' cognitive and academic performance is needed to support the introduction of standing desks in schools. It has indeed been advocated to capture such outcomes in further research, as this information is of primary importance for schools. A potential mechanism could be that standing is associated with increased energy expenditure, resulting in an effect on cognitive performance. Currently, two very small studies provide support at the proof of concept level and pilot data that standing desks might impact cognitive function positively among children or adolescents. A pilot study that explored neurocognitive benefits of standing desks in 14-year-olds across secondary schools found that the use of standing desks was associated with significant improvements in executive function and working memory capabilities over a period of about six months. The authors advocated that more research is needed, as the study was conducted in one school with no comparison group and a relatively small study sample (n = 27). Another pilot study investigated the effect of implementing standing desks for 11 weeks into a primary school classroom, and found that the intervention group significantly improved on the Digit Task Span test compared to the control group. No differences were found for the Eriksen flanker task, suggesting that standing desks are more likely to affect the short-term working memory than the inhibitory control. However no firm conclusion can be drawn from this study because its sample size was too small (n = 38) and the intervention period too short. More research is needed to provide a definitive answer.

Finally, in our previous study, only three standing desks per class were installed. The reason to choose three desks was that schools often report the high costs of standing desks as a barrier to implement them. This implied that practicable solutions need to be provided (such as installing a limited amount of desks per class) to broadly promote and disseminate the use of standing desks in schools. In addition, the financial restrictions within the project did not allow the researchers to install a large amount per class. However, this caused that pupils only stood up for 50 minutes per week on average. In the pilot study of Wick et al. who investigated the effect on cognitive function, it was recommended that using the desks for at least 1 hour per school day would be advisable to improve cognitive function. Thus, it will be important for the evaluation to install a sufficient amount of standing desks in every classroom to ensure that adolescents can stand up long enough. In the methodology of this proposal, this will be further specified.

Purpose of the study:

The primary aim of this project is to investigate the effect of implementing standing desks on adolescents' cognitive function, more specifically on memory, reasoning, verbal ability and concentration. In addition, the effect of implementing standing desks on adolescents' sitting and standing time wil be evaluated. Finally, the relationship between sleeping behavior (duration and quality) and cognitive performance will also be investigated. This will be tested via a controlled trial with a pre- and post-test design including an intervention and a control group. Providing evidence on the effect on cognitive functioning of standing desks is the first step, as it could further influence academic performances. As there is currently only preliminary evidence from studies with a small study sample and no control group, this study will definitely be of added value to the research field. In addition, if there would be strong evidence for beneficial effects, this would be a key rationale to introduce standing desks into schools and decisive factor to persuade all teachers (including the more conservative ones) to use standing desks in the classroom.

Study design:

As indicated above, the effect will be tested via a controlled trial including an intervention (3 secondary schools) and control condition (3 secondary schools). A convenience sample for the intervention group and for the control group will be selected in Flanders. The principals will be sent a recruitment letter and afterwards contacted by phone. A priori power analysis, based on a moderate effect size for cognitive function, suggests a total sample size of 90 participants (G*power 3.1.9.2; α = 0.05, 1-β = 0.80). Taking into account a response rate of 80%, the investigators will recruit about 120 adolescents (60 intervention, 60 control) to ensure that 90 participants will complete the measurements. The principals will be asked to select one class per school, with at least 20 pupils per class. In addition, it will be required that the adolescents spend a large amount of time in the same classroom (preferably at least 1/3 of lesson hours, which equals 11 lesson hours per week in the same classroom) in order to be sufficiently exposed to the desks. The investigators will inform the pupils in the classes about our study and provide an information letter for their parents. It will be specified that the standing desks will be delivered to all adolescents from a class (similar as to other health interventions that are delivered by the teacher to the entire class), but that the adolescents are free to participate in the pre- and post-test measurement. All pupils (and their parents) that agree to participate in the measurements, will first participate in the pre-test measurement (February/March 2019). Primary study outcomes will be adolescents' memory, reasoning, verbal ability and concentration (using the Cambridge Brain Science tasks). Major secondary study outcomes will be adolescents' sitting and standing time (measured by the Axivity accelerometer worn during 5 school days) on the one hand and sleep quality (using a questionnaire) and sleep duration (using Fitbits) on the other hand. Afterwards, the standing desks will be implemented for four to five months in the intervention schools (starting immediately after the pre-test). At the end of the school year (June 2019), the post-test will be conducted.*

*Due to the COVID-19 pandemic, the study was interrupted in March (after completion of the pre-test). Therefore, a new pre-test was conducted (in a new sample) in September/October 2020, which was followed by the exposure to the standing desks for approximately 4 or 5 weeks. In November/December 2020 the post-test was conducted.

Implementation of the standing desks:

To ensure that adolescents will spend sufficient time at the standing desks, 1/3 to half of the classroom will be provided with standing desks. The school will be asked to actually replace some traditional desks with these standing desks, instead of just adding standing desks to the classroom set-up to ensure as much as possible that the desks are being continuously used throughout the intervention period. Prior to installing the standing desks in the classrooms, a training session will be delivered to the teachers about the importance of using standing desks in terms of health promotion and how the teachers can motivate the pupils to use standing desks, and how the standing desks need to be safely and appropriately used. In addition, a rotation system will be suggested in which adolescents rotate every lesson hour, based on the findings and suggestions from our previous study. Further, a poster with a motivational quote will be provided to hang on the wall to remind and motivate pupils and teachers to use the desks. Finally, every month a researcher will go to the intervention class to evaluate if the standing desks are frequently used and if there are any difficulties and to encourage everyone to keep using the desks (also by providing a new poster every time). These strategies will be important, as it was found in our previous standing desk study that the use of standing desks decreased over time, probably because introducing standing desks can have a novelty effect.

Statistical analyses:

To evaluate the effect of the standing desks, Repeated Measures MANOVA will be executed with time as a within-subjects factor (pre- versus post-test) and condition as a between-subjects factor (intervention vs. control group), using MLwiN 2.31 (Centre for Multilevel Modelling, University of Bristol, UK) to take clustering of adolescents in schools into account.

ELIGIBILITY:
Inclusion Criteria:

* A 7th or 8th Grade class
* General secondary education
* Spending at least 11 lessons hours per week in one classroom

Exclusion Criteria:

* Technical or vocational secondary education

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Change in score on the 'Monkey Ladder' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing visuospatial working memory
Change in score on the 'Spatial Span' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing spatial short term memory
Change in score on the 'Token Search' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing working memory
Change in score on the 'Spatial Planning' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing planning
Change in score on the 'Digit Span' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing verbal short term memory
Change in score on the 'Double Trouble' task (Cambridge Brain Sciences test battery) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Task assessing response inhibition

SECONDARY OUTCOMES:
Change in sitting and standing time | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements. The Axivity monitor will be worn during 4 to 5 days.
  Sitting and standing time will be derived from an Axivity accelerometer that will be placed on the anterior thigh.
Change in self-reported sitting time at school (included in the questionnaire) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Children will be asked to report sitting time, using 11 response categories ranging from 'not' to 'more than 7 hours/day'.
Change in self-reported number of breaks from sitting time per school hour (included in the questionnaire) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Children will be asked to report breaks in sitting time during a normal school hour, using 7 response categories ranging from 'never' to '6 times or more'.
Change in potential determinants/correlates related to breaking up sitting time (included in the questionnaire) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Children will be asked to report their attitude towards breaking up sitting time, preference towards breaking up sitting time, self-efficacy to break up sitting time, automaticity to break up sitting time and knowledge about the advantages of breaking up sedentary time. Each correlate/potential determinant is assessed using one item on a 5-point scale ranging from 'totally disagree' to 'totally agree'. Higher scores mean a better outcome, except for the item about the self-efficacy to break up sitting time.
Sleep quality (included in the questionnaire) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Children will be asked to report the quality of their sleeping behaviour using 5 questionnaire items. Each item has 5 response categories ranging from 'never' to 'always'. The items are derived from the reliable and valid Health Behaviour in School-aged Children (HBSC)-questionnaire. Higher scores mean a worse outcome, except for the item "When I wake up in the morning, I feel rested."
Sleep quality: Waking up at night (included in the questionnaire) | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements.
  Children will be asked to report the number of breaks while sleeping (i.e. waking up at night), using 10 response categories ranging from 'never' to 'every day: more than 3 times per night'. This item is derived from the reliable and valid Health Behaviour in School-aged Children (HBSC)-questionnaire.
Sleep duration | Assessed pre-intervention and immediately after the intervention, with an average of 4 months between both measurements. The fitbit monitor will be worn during 4 to 5 days.
  Sleep duration will be derived from a fitbit monitor that will be worn on the wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté Verloigne, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: Will be published together with publication of the article(s).
Access Criteria: Dependent on journal: Probably depositing into data repositories or by publishing the data and files as supplementary information in the journal.

REFERENCES:
- [Background] Verloigne M, Ridgers ND, De Bourdeaudhuij I, Cardon G. Effect and process evaluation of implementing standing desks in primary and secondary schools in Belgium: a cluster-randomised controlled trial. Int J Behav Nutr Phys Act. 2018 Sep 27;15(1):94. doi: 10.1186/s12966-018-0726-9. PMID 30261883
- [Derived] Van Oeckel V, Deforche B, Miatton M, Poppe L, Verloigne M. Pupils' and teachers' experiences with implementing standing desks in secondary schools in Belgium. Prev Med Rep. 2025 Oct 21;60:103285. doi: 10.1016/j.pmedr.2025.103285. eCollection 2025 Dec. PMID 41209664
- [Derived] Van Oeckel V, Poppe L, Deforche B, Brondeel R, Miatton M, Verloigne M. Associations of habitual sedentary time with executive functioning and short-term memory in 7th and 8th grade adolescents. BMC Public Health. 2024 Feb 16;24(1):495. doi: 10.1186/s12889-024-18014-x. PMID 38365719
- [Derived] Verloigne M, Van Oeckel V, Brondeel R, Poppe L. Bidirectional associations between sedentary time and sleep duration among 12- to 14-year-old adolescents. BMC Public Health. 2021 Sep 15;21(1):1673. doi: 10.1186/s12889-021-11694-9. PMID 34521376